CLINICAL TRIAL: NCT05963555
Title: Evaluation of Photobiomodulation or Dry Float Therapy on Sleep Quality in Middle-aged and Elderly Individuals.
Brief Title: PBM or Dry Float Therapy on Sleep Quality in Middle-aged and Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2303738136
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-02

CONDITIONS: Sleep Quality
Keywords: Sleep Quality; Photobiomodulation; Dry Float
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Whole-Body Photobiomodulation (Experimental): Light therapy in both the visible and near-infrared range (non-UV) applied to the whole body in a light pod or bed.
  Interventions: Device: NovoThor
- Dry Float (Experimental): Simulates the effects of traditional Float-REST therapy. Instead of contact with salt water, the dry float system has a very thin membrane that cradles the body and provides a warm sensation, similar to that experienced in a traditional flotation tank.
  Interventions: Device: ZeroBody
- Localized Photobiomodulation (Experimental): Light therapy in both the visible and near-infrared range (non-UV) applied locally to only a specific body region.
  Interventions: Device: VieLight
- Control (No Intervention): Participants in the control group will be asked to keep their normal daily routine.

INTERVENTIONS:
Device: NovoThor — Following the baseline block (first four weeks), participants will use the NovoThor device 2-3 times per week for 20 minute sessions at the WVU Rockefeller Neuroscience Institute.
  Arms: Whole-Body Photobiomodulation
Device: VieLight — Following the baseline block (first four weeks), participants will use the VieLight device 2-3 times per week for 20 minute sessions and may be completed at home.
  Arms: Localized Photobiomodulation
Device: ZeroBody — Following the baseline block (first four weeks), participants will use the Zerobody device 2-3 times per week for 20 minute sessions at the WVU Rockefeller Neuroscience Institute.
  Arms: Dry Float

SUMMARY:
The main objective of this study is to assess the impact of implementing photobiomodulation (PBM) therapy, either localized or whole body, or dry float on sleep quality in middle-aged and elderly individuals experiencing sleep disturbance. As a secondary objective we will analyze the effect of the treatments on other indices of recovery (subjective and objective) via physiological monitoring in middle-aged and elderly individuals experiencing sleep disturbance.

The study will have 2 phases: Phase 1 will last 5 weeks and will serve as baseline data collection of sleep quality. Phase 2 contains the experimental conditions and will last 13 weeks. Cognitive, behavioral, and physiological tests will be done at baseline (week 1) and at the end of experimental period (week 18). Sleep tracking data will be collected daily.

DETAILED DESCRIPTION:
In summary the study participants are expected to:

* Wear a study provided smart ring (OURA Ring) through the end of the study period (at least 75% of the total study time) which measures sleep quantity/quality.
* Keep their smart phones nearby and charged while wearing their devices.
* Complete monthly surveys with questions about general well-being until the end of the study period.
* Complete a testing battery consisting of cognitive tests, behavioral and mood questionnaires, qEEG and physical assessments, in the beginning and at the end of the study period.
* Complete the designated experimental condition 2- 3x/week for 12 weeks (at least 75% of the total sessions), if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 50-85 years of age
* Able and willing to give informed consent
* No significant untreated medical history

Exclusion Criteria:

* Have no mental or physical conditions that are deemed inappropriate for study participation at investigator's discretion.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Changes in resting state electroencephalography (EEG) | Changes from baseline versus end of study week 18
  Electroencephalography (EEG) analysis looking for alterations in brain activity. A paired samples t-Test will be used to compare power activity at baseline and follow-up.
Changes in the Patient Health Questionnaire (PHQ-9) | Changes from baseline versus end of study week 18
  Participants will complete the Patient Health Questionnaire (PHQ-9) once a month. The higher the score, the more severe the symptoms of depression. Scores range from 5-9 = mild, 10-14 = moderate, 15-19 = moderate severe, 20-27 severe depression
Changes in total sleep via Oura Ring | Changes from baseline versus end of study week 18
  Oura Ring will be used to track total sleep throughout the study. Increased total sleep values will indicate better quality sleep and decrease total sleep values will indicate poorer sleep.
Changes in the Circadian Sleep Inventory | Changes from baseline versus end of study week 18
  Evaluate changes in the participants sleeping patterns. Higher values indicate poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- WVU Rockefeller Neuroscience Institute, Morgantown, West Virginia, United States